CLINICAL TRIAL: NCT00023244
Title: A Double-Blind Randomized Trial of Steroid Withdrawal in Sirolimus- and Cyclosporine-Treated Primary Transplant Recipients
Brief Title: Steroid Withdrawal in Pediatric Kidney Transplant Recipients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Effective August 13, 2004: Unanticipated high incidence of post-transplant lymphoproliferative disorder
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Cooperative Clinical Trials in Pediatric Transplantation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT SW01
Record Dates: First submitted 2001-08-29; First posted 2001-08-31 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Basiliximab; Cyclosporine; Tacrolimus; Sirolimus; Methylprednisolone; Prednisone; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroid (steroid) withdrawal (Experimental): All enrolled subjects who have not experienced an episode of acute rejection or other event resulting in removal from the study in the first 6 months after transplantation will undergo a protocol-driven biopsy at 6 months. Subjects with no clinical or histologic evidence of rejection will be eligible to be randomized and treated in a double-blinded (e.g., masked-neither subject nor health care providers will know treatment being received) fashion while continuing other immunosuppressive medications. Subjects in this arm will undergo complete steroid withdrawal by the end of 12 months post-transplant.
  Interventions: Drug: Basiliximab; Drug: Cyclosporine; Drug: Tacrolimus; Drug: Sirolimus; Drug: Methylprednisolone; Drug: Prednisone; Drug: Bactrim
- Control Treatment (Active Comparator): All enrolled subjects who have not experienced an episode of acute rejection or other event resulting in removal from the study in the first 6 months after transplantation will undergo a protocol-driven biopsy at 6 months. Subjects with no clinical or histologic evidence of rejection will be eligible to be randomized and treated in a double-blinded (e.g., masked-neither subject nor health care providers will know treatment being received) fashion while continuing other immunosuppressive medications. Subjects in this arm will be maintained on low-dose (0.15 mg/kg/day) daily steroids.
  Interventions: Drug: Basiliximab; Drug: Cyclosporine; Drug: Tacrolimus; Drug: Sirolimus; Drug: Methylprednisolone; Drug: Prednisone; Drug: Bactrim

INTERVENTIONS:
Drug: Basiliximab — Administered as a bolus intravenous injection. The first dose is given pre-operatively, the second dose is given on post-transplant day four. Dosage is determined by individual weight.
  Other Names: Simulect; Anti-CD25 monoclonal antibody, chimeric
Drug: Cyclosporine — Participants receiving cyclosporine microemulsion formula (in lieu of tacrolimus) will have the dose adjusted to maintain a whole blood trough Abbott TDx assay monoclonal level of 175-400 ng/mL (or an equivalent high pressure liquid chromatography (HPLC) level) for the first 2 weeks after transplant. The dose will subsequently be tapered to maintain a trough level of 175-300 ng/mL from week 3 to month 3, and 50-250 ng/mL from month 3 through the end of the study at month 36 (year 3).
  Other Names: CsA
Drug: Tacrolimus — Participants receiving tacrolimus (in lieu of Cyclosporine) will have the dose adjusted to maintain a whole blood trough level between 10 and 15 ng/mL for the first 4weeks after transplant. Trough levels will be maintained between 5 and 10 ng/mL thereafter throughout the duration of the study.
Drug: Sirolimus — Participants take daily (orally, either as tablets or as liquid) starting on postoperative day 1 at a dose of 6 mg/m2 and will be adjusted to maintain a trough level of 10-20 ng/mL throughout the study.
Drug: Methylprednisolone — Administered at 10 mg/kg intravenously perioperatively and on postoperative day 1.
Drug: Prednisone — Administered orally beginning on Post-Op Day 2 and maintained for all participants until day 180. Randomization will determine whether patients will maintain this treatment following day 180.
Drug: Bactrim — All subjects will receive TMP SMX (Bactrim), pneumocystis jiroveci (carinii) prophylaxis, beginning on postoperative day 1 and continuing for 6 months following transplant. Dosage: 10 mg/kg taken orally three times weekly (maximum dose 160 mg).
  Other Names: TMP SMX; trimethoprim/sulfamethoxazole

SUMMARY:
The purpose of this study is to examine the effects of withdrawing steroids on graft rejection and kidney functions in kidney transplant recipients between the ages of 0 and 20 years (prior to their 21st birthday).

Graft survival has improved in recent years in children with kidney transplants. One bad side effect of steroid maintenance therapy has been growth retardation. Doctors believe steroids might be safely withdrawn in patients that are receiving other maintenance therapies. If steroids are removed, children might catch up in their growth and also might have fewer side effects of other kinds. This study evaluates whether steroid therapy can be withdrawn in a way that does not increase graft rejection.

DETAILED DESCRIPTION:
Children receiving kidney (renal) transplantation face distressing issues in post-transplantation including but not limited to growth retardation directly attributable to corticosteroids (steroids). It is hypothesized that robust immunosuppression with sirolimus and calcineurin inhibitors (cyclosporine or tacrolimus) in conjunction with induction therapy should enable successful steroid withdrawal. A steroid-free environment could lessen side effects by enabling a child to achieve catch-up growth, reducing the need for anti-hypertensive therapy, and reducing the risk of cardiovascular disease. This trial tests the objective of providing a steroid-free state without incurring the risk of increased incidence of acute transplant rejections.

Patients are enrolled prior to kidney transplantation and receive standard evaluations. Patients receive induction therapy with basiliximab preoperatively and on Day 4 after surgery. Immunosuppressive therapy begins with sirolimus and either cyclosporine or tacrolimus on Day 1 following surgery, and with corticosteroids the day of surgery. Infection prophylaxis with Bactrim is begun on Day 1 after surgery and center-specific anti-cytomegalovirus (CMV) therapy is given for all recipients of a CMV positive kidney. At 6 months post-transplantation, all patients who have not had an episode of acute rejection undergo a renal graft biopsy. Patients who are confirmed to be free of subclinical rejection are randomized to either undergo complete steroid withdrawal or continue maintenance on daily steroids. Patients receive either steroids or placebo, while continuing other immunosuppressive medications. Patients are segregated into weight groups for steroid withdrawal that occurs over months 7 to 13. Any acute rejection event during withdrawal is confirmed by renal biopsy and managed with methylprednisolone treatment. Patients are followed for 3 years post-transplantation for analysis of growth rate, blood pressure, lipid profile and renal function as measured by serum creatinine and calculated creatinine clearances. Post-transplantation clinic visits are weekly for the first 2 months, every 2 weeks until 13 months, weekly during Month 13, every 2 weeks through Month 18, and monthly until the study ends.

Patients who exhibit evidence of acute or subclinical rejection do not continue the steroid withdrawal trial and care is managed by their pediatric renal transplant center physicians.

ELIGIBILITY:
Inclusion Criteria:

Patients may be eligible for this study if they:

* Are between the ages of 0 and 20 years (prior to their 21st birthday)
* Are receiving their first living related (e.g.,kidney from a relative or unrelated donor) or cadaver donor transplant
* Are willing to practice an acceptable method of birth control during the study, if women able to have children

Exclusion Criteria:

Patients will not be eligible for this study if they:

* Have received multiple organs
* Have received 2 or more transplants
* Have an active infection (including tuberculosis), or cancer
* Have used an experimental agent within 4 weeks of transplantation

Ages: 1 Day to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 274 (Actual)
Dates: Start 2001-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Growth, measured as change in standardized height from 6 month to 2.5 years post-transplantation | At 6 months and 2.5 years post-transplant

SECONDARY OUTCOMES:
Graft and patient survival | Throughout study
Biopsy-proven acute rejection | Throughout study
Renal function, measured by serum creatinine and the calculated creatinine clearances | Throughout study
Hypertension | Throughout study
Cushingoid features | Throughout study
Systolic and diastolic blood pressure levels | Throughout study
Fasting lipid profile | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: William Harmon, MD, Principal Investigator — Boston Children's Hospital
Locations (19):
- United States (18):
  - University of Alabama, Birmingham, Alabama
  - UCSD Medical Center, San Diego, California
  - Denver Children's Hospital, Aurora, Colorado
  - University of Florida Health Science Center, Jacksonville, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Tulane University Medical Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Children's Hospital of Boston, Boston, Massachusetts
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - The Children's Hospital of Buffalo, Buffalo, New York
  - Westchester Medical Center, Valhalla, New York
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Penn State College of Medicine, Hershey, Pennsylvania
  - LeBonheur Children's Medical Center, Memphis, Tennessee
  - Christopher Goldsbury Center, San Antonio, Texas
  - Children's Hospital and Regional Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Hospital Infantil de Mexico, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Magee JC. Steroids in pediatric kidney transplantation: a balancing act in progress. Am J Transplant. 2010 Jan;10(1):6-7. doi: 10.1111/j.1600-6143.2009.02923.x. Epub 2009 Dec 17. No abstract available. PMID 19958331
- [Background] Li L, Chang A, Naesens M, Kambham N, Waskerwitz J, Martin J, Wong C, Alexander S, Grimm P, Concepcion W, Salvatierra O, Sarwal MM. Steroid-free immunosuppression since 1999: 129 pediatric renal transplants with sustained graft and patient benefits. Am J Transplant. 2009 Jun;9(6):1362-72. doi: 10.1111/j.1600-6143.2009.02640.x. Epub 2009 May 13. PMID 19459814
- [Result] Benfield MR, Bartosh S, Ikle D, Warshaw B, Bridges N, Morrison Y, Harmon W. A randomized double-blind, placebo controlled trial of steroid withdrawal after pediatric renal transplantation. Am J Transplant. 2010 Jan;10(1):81-8. doi: 10.1111/j.1600-6143.2009.02767.x. Epub 2009 Jul 28. PMID 19663893
- [Result] McDonald RA, Smith JM, Ho M, Lindblad R, Ikle D, Grimm P, Wyatt R, Arar M, Liereman D, Bridges N, Harmon W; CCTPT Study Group. Incidence of PTLD in pediatric renal transplant recipients receiving basiliximab, calcineurin inhibitor, sirolimus and steroids. Am J Transplant. 2008 May;8(5):984-9. doi: 10.1111/j.1600-6143.2008.02167.x. PMID 18416737
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY133 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY133 — ImmPort study identifier is SDY133
- Available data/document: Study Protocol: SDY133 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY133 — ImmPort study identifier is SDY133
- Available data/document: Study summary, -design,-demographics, -files et al.: SDY133 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY133 — ImmPort study identifier is SDY133